CLINICAL TRIAL: NCT00159536
Title: Metformin Treatment of Pregnant Women With Polycystic Ovary Syndrome (PCOS)
Brief Title: Metformin in Pregnant PCOS Women
Acronym: PregMet
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PregMet
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Polycystic Ovary Syndrome
Keywords: PCOS; metformin; pregnancy; preeclampsia; diabetes; preterm delivery
MeSH Terms: conditions — Polycystic Ovary Syndrome; Pre-Eclampsia; Diabetes Mellitus; Premature Birth | interventions — Metformin; Tablets

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Metformin (Experimental): Metformin 1000mg x 2 daily
  Interventions: Drug: Metformin
- placebo (Placebo Comparator): Placebo x 2 daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Metformin — Metformin 1000 mg x 2 per day. Orally. From inclusion (before gestational week 12) to delivery. Verbal and written diet and lifestyle advices at inclusion to the study
  Other Names: metformin from Weifa 500 mg / tablet
  Arms: Metformin
Drug: Placebo — Placebo, 2 tablets x 2 daily.Orally. From inclusion (that is before gestational week 12) to delivery. Verbal and written diet and lifestyle advices at inclusion to the study
  Other Names: Placebo from Weifa
  Arms: placebo

SUMMARY:
To investigate the effect of metformin on pregnancy complications and pregnancy outcome in the II. and III. trimester of pregnancy in women with polycystic ovary syndrome.

ELIGIBILITY:
Inclusion Criteria:

* 18-45 years,
* PCOS diagnosis according to Rotterdam criteria
* single, viable, ultrasound verified fetus
* if metformin was used at conception and early pregnancy, at least 7 days of "wash out"

Exclusion Criteria:

* known liver disease or ALAT > 90 nmol/L
* known renal disease or creatinine > 110 micromol/L
* diabetes mellitus
* alcohol or drug abuse
* peroral steroid treatment
* cimetidine, anticoagulant or erythromycin treatment at time of inclusion
* not suitable for other reasons

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 257 (Actual)
Dates: Start 2005-02; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Gestational diabetes | up to delivery
incidence of metabolic syndrome and neurophysiologic parameters in offspring | Within 18 years
Preterm delivery | up to delivery
pre-eclampsia | up to delivery

SECONDARY OUTCOMES:
emesis and hyperemesis | up to delivery
Breastfeeding | One year post partum
weight change | up to delivery
blood pressure change | up to delivery
Incident of instrumental deliveries | at delivery
Hormone levels in mother and offspring | up to delivery
Snoring and sleep quality | up to delivery

CONTACTS AND LOCATIONS:
Overall Officials: Eszter I Vanky, MD, PhD, Principal Investigator — Norwegian University of Science and Technology
Locations (10):
- Norway (10):
  - Ålesund Hospital, Ålesund
  - University hospital of Bergen, Bergen
  - Central Hospital of Northern Norway, Bodø
  - Buskerud Hospital, Drammen
  - Haugesund Hospital, Haugesund
  - Ringerike Hospital, Hønefoss
  - Elvebredden Gynekologpraksis, Kristiansand
  - Lillehammer Hospital, Lillehammer
  - Stavanger University Hospital, Stavanger
  - Departments of Obstetrics and Gynecology and Endocrinology, St. Olav's Hospital, Trondheim

REFERENCES:
- [Background] Underdal MO, Stridsklev S, Oppen IH, Hogetveit K, Andersen MS, Vanky E. Does Metformin Treatment During Pregnancy Modify the Future Metabolic Profile in Women With PCOS? J Clin Endocrinol Metab. 2018 Jun 1;103(6):2408-2413. doi: 10.1210/jc.2018-00485. PMID 29659896
- [Result] Vanky E, Stridsklev S, Heimstad R, Romundstad P, Skogoy K, Kleggetveit O, Hjelle S, von Brandis P, Eikeland T, Flo K, Berg KF, Bunford G, Lund A, Bjerke C, Almas I, Berg AH, Danielson A, Lahmami G, Carlsen SM. Metformin versus placebo from first trimester to delivery in polycystic ovary syndrome: a randomized, controlled multicenter study. J Clin Endocrinol Metab. 2010 Dec;95(12):E448-55. doi: 10.1210/jc.2010-0853. Epub 2010 Oct 6. PMID 20926533
- [Result] Vanky E, Carlsen SM. Androgens and antimullerian hormone in mothers with polycystic ovary syndrome and their newborns. Fertil Steril. 2012 Feb;97(2):509-15. doi: 10.1016/j.fertnstert.2011.11.021. Epub 2011 Dec 10. PMID 22154766
- [Result] Shetelig Lovvik T, Stridsklev S, Carlsen SM, Salvesen O, Vanky E. Cervical Length and Androgens in Pregnant Women With Polycystic Ovary Syndrome: Has Metformin Any Effect? J Clin Endocrinol Metab. 2016 Jun;101(6):2325-31. doi: 10.1210/jc.2015-3498. Epub 2016 Feb 2. PMID 26835542
- [Result] Hanem LGE, Stridsklev S, Juliusson PB, Salvesen O, Roelants M, Carlsen SM, Odegard R, Vanky E. Metformin Use in PCOS Pregnancies Increases the Risk of Offspring Overweight at 4 Years of Age: Follow-Up of Two RCTs. J Clin Endocrinol Metab. 2018 Apr 1;103(4):1612-1621. doi: 10.1210/jc.2017-02419. PMID 29490031
- [Result] Hanem LGE, Salvesen O, Juliusson PB, Carlsen SM, Nossum MCF, Vaage MO, Odegard R, Vanky E. Intrauterine metformin exposure and offspring cardiometabolic risk factors (PedMet study): a 5-10 year follow-up of the PregMet randomised controlled trial. Lancet Child Adolesc Health. 2019 Mar;3(3):166-174. doi: 10.1016/S2352-4642(18)30385-7. Epub 2019 Jan 29. PMID 30704873
- [Derived] Ryssdal M, Skage JE, Jarmund AH, Hanem LGE, Lovvik TS, Giskeodegard GF, Iversen AC, Vanky E. Metformin Treatment in PCOS Pregnancies Reduces Maternal Infections and Increases the Risk of Allergies and Eczema in the Offspring: Post Hoc Analyses of Two Randomised Controlled Trials and One Follow-Up Study. BJOG. 2025 Nov;132(12):1823-1832. doi: 10.1111/1471-0528.18320. Epub 2025 Aug 11. PMID 40785326
- [Derived] Ujvari D, Trouva A, Hirschberg AL, Vanky E. Maternal serum levels of prokineticin-1 related to pregnancy complications and metformin use in women with polycystic ovary syndrome: a post hoc analysis of two prospective, randomised, placebo-controlled trials. BMJ Open. 2023 Nov 21;13(11):e073619. doi: 10.1136/bmjopen-2023-073619. PMID 37989369
- [Derived] Trouva A, Alvarsson M, Calissendorff J, Asvold BO, Vanky E, Hirschberg AL. Thyroid Status During Pregnancy in Women With Polycystic Ovary Syndrome and the Effect of Metformin. Front Endocrinol (Lausanne). 2022 Feb 21;13:772801. doi: 10.3389/fendo.2022.772801. eCollection 2022. PMID 35265033
- [Derived] Stokkeland LMT, Giskeodegard GF, Ryssdal M, Jarmund AH, Steinkjer B, Madssen TS, Stafne SN, Stridsklev S, Lovvik TS, Iversen AC, Vanky E. Changes in Serum Cytokines Throughout Pregnancy in Women With Polycystic Ovary Syndrome. J Clin Endocrinol Metab. 2022 Jan 1;107(1):39-52. doi: 10.1210/clinem/dgab684. PMID 34529073
- [Derived] Andrae F, Abbott D, Stridsklev S, Schmedes AV, Odsaeter IH, Vanky E, Salvesen O. Sustained Maternal Hyperandrogenism During PCOS Pregnancy Reduced by Metformin in Non-obese Women Carrying a Male Fetus. J Clin Endocrinol Metab. 2020 Dec 1;105(12):3762-70. doi: 10.1210/clinem/dgaa605. PMID 32866967
- [Derived] Greger HK, Hanem LGE, Ostgard HF, Vanky E. Cognitive function in metformin exposed children, born to mothers with PCOS - follow-up of an RCT. BMC Pediatr. 2020 Feb 10;20(1):60. doi: 10.1186/s12887-020-1960-2. PMID 32039724
- [Derived] Underdal MO, Salvesen O, Henriksen AH, Andersen M, Vanky E. Impaired Respiratory Function in Women With PCOS Compared With Matched Controls From a Population-Based Study. J Clin Endocrinol Metab. 2020 Jan 1;105(1):dgz053. doi: 10.1210/clinem/dgz053. PMID 31613965
- [Derived] Stridsklev S, Salvesen O, Salvesen KA, Carlsen SM, Vanky E. Uterine Artery Doppler in Pregnancy: Women with PCOS Compared to Healthy Controls. Int J Endocrinol. 2018 Aug 16;2018:2604064. doi: 10.1155/2018/2604064. eCollection 2018. PMID 30186323
- [Derived] Hjorth-Hansen A, Salvesen O, Engen Hanem LG, Eggebo T, Salvesen KA, Vanky E, Odegard R. Fetal Growth and Birth Anthropometrics in Metformin-Exposed Offspring Born to Mothers With PCOS. J Clin Endocrinol Metab. 2018 Feb 1;103(2):740-747. doi: 10.1210/jc.2017-01191. PMID 29165598
- [Derived] Christiansen SC, Vanky E, Klungland H, Stafne SN, Morkved S, Salvesen KA, Saether M, Carlsen SM. The effect of exercise and metformin treatment on circulating free DNA in pregnancy. Placenta. 2014 Dec;35(12):989-93. doi: 10.1016/j.placenta.2014.09.010. Epub 2014 Sep 23. PMID 25282112
- [Derived] Helseth R, Vanky E, Stridsklev S, Vogt C, Carlsen SM. Maternal and fetal insulin levels at birth in women with polycystic ovary syndrome: data from a randomized controlled study on metformin. Eur J Endocrinol. 2014 Apr 10;170(5):769-75. doi: 10.1530/EJE-13-0859. Print 2014 May. PMID 24595965
- [Derived] Carlsen SM, Martinussen MP, Vanky E. Metformin's effect on first-year weight gain: a follow-up study. Pediatrics. 2012 Nov;130(5):e1222-6. doi: 10.1542/peds.2012-0346. Epub 2012 Oct 15. PMID 23071212